CLINICAL TRIAL: NCT05098236
Title: Effect of Visual Retraining on Visual Loss Following Visual Cortical Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Krystel Huxlin, Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000075; R01EY027314 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-10-28 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Vision Loss Partial; Hemianopia; Hemianopia Homonymous; Quadrantanopia; Stroke, Ischemic
MeSH Terms: conditions — Hemianopsia; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cortically Blind Subjects (Experimental)
  Interventions: Other: Training in the Blind Field
- Control (Placebo Comparator)
  Interventions: Other: Training in the Sighted Field

INTERVENTIONS:
Other: Training in the Blind Field — A computer software and chin-rest necessary to perform visual training will be loaned to each subject to be used at home. Subjects will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion, the presence of motion, or the orientation of a visual stimulus (either a small cloud of dots or bars) located at a predetermined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. Subjects will train daily (about 40-60 minutes total), 5 to 7 days per week for at least 3 and up to 12 months at a time.
  Arms: Cortically Blind Subjects
Other: Training in the Sighted Field — This training will take place in lab at the University of Rochester Medical Center. Subject will perform one daily training session, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion, the presence of motion, or the orientation of a visual stimulus (either a small cloud of dots or bars) located at a predetermined location in the visual field. The computer program will automatically create a record of patient performance during each training session. Subjects will train daily (about 30-40 minutes total), 5 to 7 days per week for at 7 - 14 days.
  Arms: Control

SUMMARY:
This project is intended to collect data using standard clinical tests and psychophysics to quantify the effect of visual cortical damage on the structure of the residual visual system, visual perception, spatial awareness, and brain function. The investigators will also assess the effect of intensive visual retraining on the residual visual system, processing of visual information and the use of such information in real-world situations following damage. This research is intended to improve our understanding of the consequences of permanent visual system damage in humans, of methods that can be used to reverse visual loss, and of brain mechanisms by which visual recovery is achieved.

ELIGIBILITY:
Cortically Blind Subject Inclusion Criteria:

* Subjects between the ages of 17 and 75, who have sustained damage to primary visual cortex at age 17 or later, and are rendered blind over a portion of their visual field.
* Subjects must have some intact visual cortical areas (other than primary visual cortex) in the damaged brain hemisphere. This assessment will be made from MRI or CT scans of the subject's head, which will be obtained via standard release from their neurologist.
* Subjects who demonstrate a clear deficit in either simple or complex visual perception in portions of their visual field.
* Subjects who are competent and responsible, as determined by the Principal Investigator.
* Subjects who will receive retinal electrophysiology (mfERG) testing must have a report from their ophthalmologist stating that they are able to receive dilating drops

Cortically Blind Subject Exclusion Criteria:

* Subjects who do not possess damage of primary visual cortex or its immediate afferents
* Subjects who are suffering from an active disease process involving their nervous system.
* Subjects who are unable to fixate visual targets precisely with their eyes
* Subjects who have unreliable vision fields from prior testing indicated by greater than 20% fixation losses, false positives or false negatives
* Best corrected visual acuity worse than 20/40 in either eye
* Impaired foveal sensitivity as indicated by visual field tests
* Presence of vision loss from ocular disease or disorder
* Presence of bilateral visual acuity loss from any source
* Subjects who are suffering from one-sided attentional neglect
* Subjects who have impaired auditory thresholds that would influence test results and training efficacy (all our testing and training involves sound as a cue for trial/stimulus onset or as feedback)
* Persons who lack the competence or are otherwise unable to perform the visual training exercises as directed.

Control Subject Inclusion Criteria:

* Subjects must be between the ages of 17 and 75 years of age
* Subjects must report no history of neurological disorder.
* Subjects who are competent and responsible, as determined by the Principal Investigator.

Control Subject Exclusion criteria:

* Subjects who possess damage to the visual system
* Subjects who are suffering from an active disease process involving their nervous system.
* Subjects who are unable to fixate visual targets precisely with their eyes
* Best corrected visual acuity worse than 20/40 in either eye
* Presence of vision loss from ocular disease or disorder
* Presence of bilateral visual acuity loss from any source
* Subjects who are suffering from one-sided attentional neglect
* Subjects who have impaired auditory thresholds that would influence test results and training efficacy (all our testing and training involves sound as a cue for trial/stimulus onset or as feedback)
* Persons who lack the competence or are otherwise unable to perform the visual testing/training exercises as directed.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2003-09-26 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Direction Discrimination Threshold | Baseline, 4-months, 12-months
  For each subject, the investigators will measure the change in ability to detect differences in the motion direction of visual stimuli relative to horizontal, measured in degrees of visual angle. These assessments will be based on what can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.
Direction Integration Threshold | Baseline to 4-months, 12-months
  This will measure the change in ability of subjects to integrate across a range of motion directions measured in degrees of visual angle. These assessments will be based on what range of motion directions can be reliably integrated at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.
Contrast Sensitivity for Direction | Baseline, 4-months, 12-months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for direction discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the motion direction of visual stimuli that are also varying in contrast against a grey background. We will measure the luminance contrast that can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.
Contrast Sensitivity for Static Orientation | Baseline, 4-months, 12-months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for static orientation discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the orientation of non-moving visual stimuli that vary in contrast against a grey background. We will measure the luminance that can be reliably detected at a 72-75% correct level of performance.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.

SECONDARY OUTCOMES:
Humphrey 10-2 and 24-2 perimetry | Baseline, 4-months, 12-months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.
Goldmann perimetry | Baseline, 4-months, 12-months
  The investigators will measure the change in area of vision (degrees squared) as encompassed by each isopter, measured by one of 3 different light stimuli.
  The 3 isopters which will be compared are:
  I2e 1asb, 0.25 mm^2 I4e 10asb, 0.25 mm^2 V4e 1000asb, 64 mm^2
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.
MAIA Visual Field Perimetry | Baseline, 4-months, 12-months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-months, then baseline to 12-months from start of training.

CONTACTS AND LOCATIONS:
Locations (1):
- Flaum Eye Institute, University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No